CLINICAL TRIAL: NCT04395053
Title: Pharmacokinetic Evaluation Study of Healthy Chinese Volunteers After Oral Administration of SHR1459 Tablets in Old and New Formulation
Brief Title: A Bioavailability Study of SHR1459 on Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SHR1459-I-104
Record Dates: First submitted 2020-04-10; First posted 2020-05-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-07

CONDITIONS: Healthy Adult Subjects
Keywords: Bioavailability evaluation; Old formulation; New formulation

STUDY DESIGN:
Intervention Model Description: * Experimental: Treatment group TR Intervention: Drug: SHR1459, new formulation; Intervention: Drug: SHR1459, old formulation.
  * Experimental: Treatment group RT Intervention: Drug: SHR1459, old formulation; Intervention: Drug: SHR1459, new formulation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group TR (Experimental): Intervention: Drug: SHR1459, new formulation; Intervention: Drug: SHR1459, old formulation.
  Interventions: Drug: SHR1459
- Treatment group RT (Experimental): Intervention: Drug: SHR1459, old formulation; Intervention: Drug: SHR1459, new formulation.
  Interventions: Drug: SHR1459

INTERVENTIONS:
Drug: SHR1459 — TR group:
  The first period，the subjects will be administrated with SHR-1459 in new formulation, then conduct blood collection within 48h; 7 days washout； The second period，the subjects will be administrated with SHR-1459 in old formulation, then conduct blood collection within 48h.
  RT group:
  The first period，the subjects will be administrated with SHR-1459 in old formulation, then conduct blood collection within 48h; 7 days washout； The second period，the subjects will be administrated with SHR-1459 in new formulation, then conduct blood collection within 48h.
  Other Names: BTK inhibitor

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics of healthy Chinese volunteers after oral administration of SHR1459 tablets in new and old formulations.

The secondary objective of the study is to evaluate the safety after single dose of SHR1459 orally in healthy Chinese subjects.

DETAILED DESCRIPTION:
The PK parameters (AUC0-t, AUC0-inf, Cmax, Tmax, T1/2z, CL/F and Vz/F etc.) will be calculated to evaluate the pharmacokinetics of healthy Chinese volunteers after oral administration of SHR1459 tablets in new and old formulations.

During the study, the safety will be assessed by vital signs, physical examination, laboratory examination (hematology, blood biochemistry, urinalysis, coagulation examination), 12-lead electrocardiogram. The incidence and severity degree of adverse events and severe adverse events will be evaluated based on CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged 18 or above (including 18 years old) at the date of signing the informed consent;
2. Body weight ≥ 50kg, body mass index (BMI) within the range of 19 ~ 26kg /m2 (including 19 and 26 kg/m2) (BMI= weight (kg)/height 2 (m2));
3. The subjects were able to communicate well with the researchers, understand and comply with the requirements of this study, understand and sign the informed consent;
4. Consent to abstinence or take effective non-drug contraception measures during the study and for at least 3 months after the last drug administration.

Exclusion Criteria:

1. Anyone who has suffered from any clinical serious disease such as the circulatory system, endocrine system, nervous system, digestive system, respiratory system, urogenital system, hematology, immunology, psychiatry and metabolic abnormalities, or any other disease which can affect the study results. Researchers should focus on the following medical history: inflammatory gastroenteritis, gastroesophageal reflux, gastrointestinal or rectal bleeding, history of pancreatic injury or pancreatitis; larger history of surgery such as gastrectomy, gastrointestinal anastomosis or bowel resection;
2. Have a history of allergies to drugs, food or other substances;
3. Those who have undergone surgery within 4 weeks before the trial, or plan to undergo surgery during the study period;
4. Those who have taken any drug (including Chinese herbal medicine, vitamins, calcium tablets and other food supplements) within 14 days before the study; Those who have taken any drug that inhibits or induces liver metabolic enzymes within 30 days before the study (such as inducer-barbiturate carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors-SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative hypnotics, vera pamil, fluoroquinolones, antihistamines);
5. Those who participated in any clinical trial and took any clinical trial drugs within 3 months before the trial;
6. Those who donated blood or suffered heavy blood loss (≥200 mL), received blood transfusions, or used blood products within 3 months before enrollment;
7. Volunteers who cannot adopt one or more non-drug contraception measures during the trial;
8. Those who have special requirements on diet and cannot follow a unified diet;
9. The subjects refused to stop any beverage or food containing methylxanthine, such as coffee, tea, cola, chocolate, etc. within 48 hours before the first dose until the end of the study; the subjects refused to discontinue any beverage or food containing grapefruit within 7 days before the first dose until the end of the study;
10. Smokers or those who smoked more than 5 cigarettes per day in the 3 months before the trial or who could not stop using any tobacco products during the trial;
11. Alcoholics or frequent drinkers within 6 months before the trial, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of 40% spirits or 150 mL of wine), or those who receive the breath alcohol test and the results are positive, or who cannot stop using any alcoholic products during the trial;
12. Those who receive the drug abuse or urine drug screening test and the results are positive.
13. Those who regularly use sedatives, sleeping pills or other addictive drugs, have used soft drugs (such as cannabis) within 3 months before the trial or hard drugs (such as cocaine, phencyclidine, etc.) within 1 year before the trial;
14. Those with abnormal vital signs (systolic blood pressure < 90 mmHg or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg; heart rate < 55 bpm or > 100 bpm) or the results of various clinical laboratory examination (including physical examination, electrocardiogram, chest radiograph, cardiac ultrasound, hematology, blood biochemistry, urinalysis, coagulation examination and virus serological detection) are abnormal and clinically significant based on the judgment of the clinical researchers;
15. Creatinine clearance (CLCr) < 80 mL/min, creatinine clearance should be calculated using the standard Cockcroft-Gault formula;
16. Volunteers are not able to complete the study for other reasons or other factors that are not suitable for participating in the study, as judged by the researchers.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-28 (Actual); Primary Completion 2020-07-11 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameter: Cmax of SHR1459 | through study completion, an average of 29 days
  Peak plasma concentration （Cmax）of SHR1459
Pharmacokinetics parameter: AUC of SHR1459 | through study completion, an average of 29 days
  Area under the plasma concentration versus time curve （AUC）of SHR1459

SECONDARY OUTCOMES:
Pharmacokinetics parameter: Tmax of SHR1459 | through study completion, an average of 29 days
  Time of maximum observed concentration (Tmax) of SHR1459
Pharmacokinetics parameter: T1/2z of SHR1459 | through study completion, an average of 29 days
  Half time (T1/2z) of SHR1459
Pharmacokinetics parameter: CL/F of SHR1459 | through study completion, an average of 29 days
  Total body clearance for extravascular administration (CL/F) of SHR1459
Pharmacokinetics parameter: Vz/F of SHR1459 | through study completion, an average of 29 days
  Volume of distribution (Vz/F) of SHR1459
The number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | through study completion, an average of 29 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China